CLINICAL TRIAL: NCT07332728
Title: Prospective Observational Evaluation of the Association Between Perioperative Changes in Diaphragmatic Excursion and Postoperative Oxygenation and Hypoxemia in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Diaphragmatic Excursion Changes and Postoperative Oxygenation After Laparoscopic Cholecystectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Haseki Training and Research Hospital
Other Study IDs: serpil Diaphragm US
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Perioperative Diaphragmatic Excursion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard perioperative care with observational diaphragm ultrasonography — No therapeutic intervention is applied in this study. All patients receive standard perioperative anesthesia and surgical care according to institutional routine. Diaphragmatic excursion is assessed non-invasively using ultrasonography in the preoperative period and at 15 minutes postoperatively in the post-anesthesia care unit. Oxygenation parameters and respiratory variables are recorded for observational analysis only.

SUMMARY:
Laparoscopic cholecystectomy and the associated pneumoperitoneum can impair diaphragmatic mechanics and reduce postoperative oxygenation. This prospective observational study aims to evaluate perioperative changes in diaphragmatic excursion measured by ultrasonography and to investigate their association with early postoperative oxygenation parameters and hypoxemia. By correlating diaphragmatic excursion changes with SpO₂/FiO₂ and the ROX index, the study seeks to clarify the physiological contribution of diaphragmatic dysfunction to postoperative hypoxemia in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years
* Scheduled for elective laparoscopic cholecystectomy under general anesthesia
* Able to undergo diaphragm ultrasonography (no preoperative barrier to assessment)
* Able to cooperate with preoperative and early postoperative diaphragm measurements
* Postoperative oxygenation data available (SpO₂, FiO₂, and SpO₂/FiO₂ can be recorded)
* Provided written informed consent

Exclusion Criteria:

* Morbid obesity (BMI ≥ 40 kg/m²)
* Known diaphragmatic paralysis, phrenic nerve injury, or hemidiaphragm dysfunction
* Severe COPD, restrictive lung disease, or advanced parenchymal lung disease
* Preoperative home oxygen therapy or CPAP/BiPAP/home mechanical ventilation
* Conversion to open surgery (laparoscopic → open)
* Hemodynamic instability preoperatively or intraoperatively; emergency/complicated surgery
* Factors preventing ultrasound assessment (e.g., marked upper abdominal gas, large scar/wound, severe subcutaneous edema)
* Same-day discharge cases with <24-hour observation
* Inability to complete measurements (e.g., severe cognitive impairment, poor cooperation, severe pain preventing measurement)
* Incomplete data not compatible with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18-75 years undergoing elective laparoscopic cholecystectomy under general anesthesia at a tertiary care center. Eligible participants are patients without known diaphragmatic dysfunction or severe underlying pulmonary disease, in whom perioperative diaphragm ultrasonography and postoperative oxygenation measurements can be reliably performed. All participants provide written informed consent and receive standard perioperative care without any study-related intervention.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
diaphragmatic excursion (ΔDE) and postoperative hypoxemia | Preoperative baseline and 15 minutes after admission to the post-anesthesia care unit (PACU).
  Association between perioperative change in diaphragmatic excursion (ΔDE) and postoperative hypoxemia, defined as SpO₂ < 92% and/or a clinically significant decrease in the SpO₂/FiO₂ ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Result] Rustagi PS, Yadav A, Nellore SS. Ultrasonographic evaluation of diaphragmatic excursion changes after major laparoscopic surgeries in the Trendelenburg position under general anaesthesia: A prospective observational study. Indian J Anaesth. 2023 Nov;67(Suppl 4):S274-S280. doi: 10.4103/ija.ija_643_23. Epub 2023 Nov 21. PMID 38187984
- [Result] Yao XY, Li HM, Sun BW, Zhang YY, Feng JG, Jia J, Liu L. Ultrasound assessment of diaphragmatic dysfunction in non-critically ill patients: relevant indicators and update. Front Med (Lausanne). 2024 Jun 18;11:1389040. doi: 10.3389/fmed.2024.1389040. eCollection 2024. PMID 38957305
- [Result] Yan T, Yu Q, Li CQ, Xu ZZ, Ma JH, Xie M, Zhu SN, Wang DX, Li SL. Maximal inspiratory diaphragmatic ultrasound predicts postoperative pulmonary complications after upper abdominal surgery. Ann Intensive Care. 2025 Aug 18;15(1):121. doi: 10.1186/s13613-025-01531-2. PMID 40824343